CLINICAL TRIAL: NCT00522509
Title: Preoperative Hepatic Arterial Infusion Chemotherapy in Patients Undergoing Liver Resection for Colorectal Liver Metastases
Brief Title: Preoperative Hepatic Arterial Infusion Chemotherapy
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: IRCCS San Raffaele (Other)
Other Study IDs: Neoadjuvant HAIC
Record Dates: First submitted 2007-08-28; First posted 2007-08-29 (Estimated); Last update posted 2007-08-29 (Estimated); Status verified 2007-05

CONDITIONS: Colorectal Liver Metastases
MeSH Terms: interventions — Floxuridine

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Retrospective

INTERVENTIONS:
Drug: Floxuridine FUDR

SUMMARY:
To assess the feasibility and results of liver resection after preoperative hepatic artery infusion (HAI) chemotherapy with FUDR.

DETAILED DESCRIPTION:
Between 1995 and 2004, 239 patients with isolated colorectal liver metastases received HAI chemotherapy with neoadjuvant intent. Fifty of these patients underwent subsequent curative liver resection (HAI group).

Postoperative morbidity, liver function tests, and long term outcomes were evaluated. Adverse events related to HAI chemotherapy were also evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable liver metastases
* Potentially resectable liver metastases

Exclusion Criteria:

* Extrahepatic disease

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1995-12

CONTACTS AND LOCATIONS:
Overall Officials: Luca Aldrighetti, M.D, PhD, Principal Investigator — Department of Surgery - Liver Unit, Scientific Institute San Raffaele,
Locations (1):
- Department of Surgery - Liver Unit, Scientific Institute San Raffaele,, Milan, Italy